CLINICAL TRIAL: NCT00818883
Title: A Phase 3, Double-Blind, Randomized, Efficacy and Safety Study of the TAK 491 Plus Chlorthalidone Fixed-Dose Combination Compared With TAK-491 and Hydrochlorothiazide Coadministration Therapy in Subjects With Moderate to Severe Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil and Chlorthalidone in Participants With Moderate to Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491CLD_306; U1111-1112-7119 (Registry Identifier: WHO)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Hypertensive; Blood Pressure, High; Vascular Disease; Cardiovascular Disease; Drug Therapy
MeSH Terms: conditions — Essential Hypertension; Hypertension; Vascular Diseases; Cardiovascular Diseases | interventions — azilsartan medoxomil; Chlorthalidone; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and hydrochlorothiazide

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablet, orally, once daily and hydrochlorothiazide placebo-matching tablets, orally, once daily for up to 10 weeks.
  For participants who do not achieve target blood pressure by Week 6, the dose of chlorthalidone will be increased for the remaining 4 weeks of treatment.
  Other Names: TAK-491; TAK-491CLD
  Arms: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD
Drug: Azilsartan medoxomil and hydrochlorothiazide — Azilsartan medoxomil 40 mg, tablets, orally, once daily and hydrochlorothiazide 12.5 mg, tablets, orally, once daily for up to 10 weeks.
  For participants who do not achieve target blood pressure by Week 6, the dose of hydrochlorothiazide will be increased for the remaining 4 weeks of treatment.
  Other Names: TAK-491; TAK-491CLD
  Arms: Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD

SUMMARY:
The purpose of this study is to compare the antihypertensive effect of chlorthalidone vs hydrochlorothiazide when each is used with azilsartan medoxomil, once daily (QD), in participants with moderate to severe essential hypertension.

DETAILED DESCRIPTION:
According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive agents, hypertension remains inadequately controlled; only about one-third of patients continue to maintain control successfully.

Although most antihypertensive agents are effective at the appropriate dose, the majority have side effects that limit their use. As a class, angiotensin II receptor blockers generally are considered more tolerable than other classes of antihypertensive agents. TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker being evaluated by Takeda to treat essential hypertension.

Treatments for essential hypertension commonly include use of a thiazide-like diuretic, either alone or as part of combination treatment. Although chlorthalidone was commonly prescribed in the past, its use has widely been replaced with hydrochlorothiazide, presumably due to a lack of available combination products containing chlorthalidone, the assumption that hydrochlorothiazide and chlorthalidone have similar antihypertensive effects and cardiovascular benefits, and the perception that chlorthalidone use is associated with a greater frequency of hypokalemia. However, the frequency of hypokalemia with chlorthalidone use is relatively low in the dose range of 12.5 to 25 mg and these doses have been shown to be associated with potent blood pressure reduction. Several long-term outcomes trials have shown that blood pressure reductions associated with chlorthalidone treatment reduce risk of cardiovascular morbidity and mortality.

Most hypertensive patients require two or more agents to achieve target blood pressure and diuretics are commonly used in combination with other antihypertensive agents. This trial is designed to compare chlorthalidone and hydrochlorothiazide when coadministered with azilsartan medoxomil.

Participants in this study will receive either chlorthalidone or hydrochlorothiazide in combination with azilsartan medoxomil. Total commitment time for this study is about 13 weeks. Participants will be required to wear a blood pressure monitor for three 24 hours periods during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Is treated with antihypertensive therapy and has a post-washout mean sitting clinic SBP greater than or equal to 160 and less than or equal to 190 mm Hg on Day -1; or the participant has not received antihypertensive treatment within 28 days prior to Screening and has a mean sitting clinic SBP greater than or equal to 160 and less than or equal to 190 mm Hg at the Screening Visit and on Day -1.
2. Females of childbearing potential who are sexually active agree to routinely use adequate contraception from Screening through 30 days after the last administered study drug dose.
3. Has clinical laboratory test results (clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or the investigator does not consider the results to be clinically significant.
4. Is willing to discontinue current antihypertensive medications on Day -21 or Day -28 if the participant is on amlodipine or chlorthalidone.

Exclusion Criteria:

1. Has a mean sitting clinic diastolic blood pressure greater than 119 mm Hg on Day -1.
2. Has a baseline 24-hour ambulatory blood pressure monitoring reading of insufficient quality.
3. Works a night (third) shift (defined as 11 PM [2300] to 7 AM [0700]).
4. Has an upper arm circumference less than 24 cm or greater than 42 cm.
5. Is noncompliant (less than 70% or greater than 130%) with study medication during the placebo run-in period.
6. Has secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
7. Has a recent history (within the last 6 months) of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
8. Has clinically significant cardiac conduction defects (ie, third-degree atrioventricular block, sick sinus syndrome, atrial fibrillation, or atrial flutter).
9. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
10. Has severe renal dysfunction or disease [based on estimated glomerular filtration rate less than 30 mL/min/1.73m2 at Screening].
11. Has known or suspected unilateral or bilateral renal artery stenosis.
12. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those participants with basal cell or stage I squamous cell carcinoma of the skin).
13. Has poorly-controlled type 1 or type 2 diabetes mellitus at Screening.
14. Has hypokalemia or hyperkalemia (defined as serum potassium outside of the normal reference range of the central laboratory).
15. Has an alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
16. Has any other known serious disease or condition that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
17. Has known hypersensitivity to angiotensin II receptor blockers or thiazide-type diuretics or other sulfonamide-derived compounds.
18. Has been randomized in a previous azilsartan medoxomil study.
19. Currently participating in another investigational study or is receiving or has received any investigational compound within 30 days prior to Screening.
20. Has a history of drug abuse or a history of alcohol abuse within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Takeda
Locations (53):
- United States (50):
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Scottsboro, Alabama
  - Gilbert, Arizona
  - Sierra Vista, Arizona
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Wheat Ridge, Colorado
  - Milford, Connecticut
  - Adventura, Florida
  - Aventura, Florida
  - Brooksville, Florida
  - Crystal River, Florida
  - DeLand, Florida
  - Doral, Florida
  - Miami, Florida
  - Naranja, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Stockbridge, Georgia
  - Suwanee, Georgia
  - Huntsville, Illinois
  - Bloomington, Indiana
  - Valparaiso, Indiana
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - West Yarmouth, Massachusetts
  - Ann Arbor, Michigan
  - City of Saint Peters, Missouri
  - St Louis, Missouri
  - New Windsor, New York
  - Asheboro, North Carolina
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Downingtown, Pennsylvania
  - Lancaster, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Goose Creek, South Carolina
  - Taylors, South Carolina
  - Bryan, Texas
  - San Antonio, Texas
  - Ettrick, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Russia (3):
  - Moscow
  - Perm
  - Saint Petersburg

REFERENCES:
- [Derived] Bakris GL, Sica D, White WB, Cushman WC, Weber MA, Handley A, Song E, Kupfer S. Antihypertensive efficacy of hydrochlorothiazide vs chlorthalidone combined with azilsartan medoxomil. Am J Med. 2012 Dec;125(12):1229.e1-1229.e10. doi: 10.1016/j.amjmed.2012.05.023. Epub 2012 Aug 30. PMID 22939358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 66 investigative sites in the Russian Federation and the United States from 20 January 2009 to 30 November 2009.
Pre-assignment Details: Participants with patients with moderate to severe essential hypertension were enrolled in one of 2, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD: Azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablet, orally, once daily and hydrochlorothiazide placebo-matching tablets, orally, once daily for up to 10 weeks.
  For participants who do not achieve target blood pressure by Week 6, the dose of chlorthalidone will be increased for the remaining 4 weeks of treatment.
- Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD: Azilsartan medoxomil 40 mg, tablets, orally, once daily and hydrochlorothiazide 12.5 mg, tablets, orally, once daily for up to 10 weeks.
  For participants who do not achieve target blood pressure by Week 6, the dose of hydrochlorothiazide will be increased for the remaining 4 weeks of treatment.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Started | 303 | 306
Completed | 252 | 260
Not Completed | 51 | 46
Not completed — Adverse Event | 28 | 19
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 16 | 14
Not completed — Lack of Efficacy | 0 | 2
Not completed — Other | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD | Total
Number analyzed (Participants) | 303 | 306 | 609
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.79) | 55.9 (10.97) | 56.4 (10.88)
Age, Customized [Number; unit: participants]
  <45 years | 43 | 50 | 93
  Between 45 and 64 years | 189 | 195 | 384
  ≥65 years | 71 | 61 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 155 | 313
  Male | 145 | 151 | 296
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 28 | 68
  Not Hispanic or Latino | 173 | 184 | 357
  Unknown or Not Reported | 90 | 94 | 184
Race (NIH/OMB) [Number; unit: participants] — Participants could choose more than 1 category for race. Participants who indicated more than 1 race category are included in each category indicated, and they are also included in the multiracial category. Thus, the sum of the number of participants by racial category may be greater than the total number of participants in the treatment group.
  participants
    American Indian or Alaska Native | 6 | 1 | 7
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 46 | 38 | 84
    White | 252 | 265 | 517
    More than one race | 5 | 0 | 5
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 213 | 214 | 427
  Russian Federation | 90 | 92 | 182
Estimated glomerular filtration rate (eGFR) [Number; unit: participants] — eGFR based on calculated creatinine clearance.
  Categories:
  Normal renal function (≥90 mL/min/1.73 m2); Mild renal impairment(≥60 to <90 mL/min/1.73 m2); Moderate renal impairment (≥30 to <60 mL/min/1.73 m2)
  participants
    Moderate impairment | 23 | 24 | 47
    Mild impairment | 180 | 184 | 364
    Normal | 100 | 98 | 198
Weight [Mean (Standard Deviation); unit: kg] | 87.60 (19.181) | 90.61 (19.252) | 89.11 (19.260)
Height [Mean (Standard Deviation); unit: cm] | 168.9 (10.08) | 168.8 (9.69) | 168.9 (9.88)
Body Mass Index (BMI) [Median (Standard Deviation); unit: kg/m2] | 30.7 (6.12) | 31.8 (6.10) | 31.2 (6.13)
Chronic Kidney Disease (CKD) Status [Number; unit: participants] — Participant was considered to have CKD if their eGFR was <60 ml/min/1.73 m2 or urinary albumin:creatinine ratio was >200 mg albumin/g creatinine at Screening.
  Includes all randomized participants.
  participants | 24 | 24 | 48
Diabetes status [Number; unit: participants] | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough, Sitting, Clinic Systolic Blood Pressure
Description: The change in sitting trough clinic systolic blood pressure measured at each week indicated including final visit relative to baseline. Systolic blood pressure is the average of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline, Week 6 and Week 10.
Population: Full analysis set, defined as all randomized participants who received at least 1 dose of active single-blind or double-blind study medication, with both a baseline value and at least 1 value during the treatment period, with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=295; n=292) | -35.1 (0.97) | -29.5 (0.98)
  Week 10 (n=295; n=292) | -37.8 (0.91) | -32.8 (0.91)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; Analysis of Covariance (ANCOVA) model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 6 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Overall type I error rate controlled using stepwise testing procedure. First treatment test done at Week 6. If statistically significant at significance level of 5%, then treatment comparison at Week 10 was performed. Tested at 5% significance level; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-8.3 to -2.9]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 10 data; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.0, 95% CI [-7.5 to -2.5]

2. Secondary Outcome: Change From Baseline in Trough, Sitting, Clinic Diastolic Blood Pressure
Description: The change in sitting trough clinic diastolic blood pressure measured at each week indicated including final visit relative to baseline. Diastolic blood pressure is the average of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=295; n=292) | -15.0 (0.55) | -11.2 (0.55)
  Week 10 (n=295; n=292) | -16.4 (0.50) | -13.7 (0.51)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 6 data; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-5.2 to -2.2]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 10 data; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-4.1 to -1.3]

3. Secondary Outcome: Change From Baseline in Mean Trough Systolic Blood Pressure (22 to 24 Hours After Dosing) as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough systolic blood pressure measured at each week indicated including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179, n=162) | -25.7 (1.11) | -18.4 (1.16)
  Week 10 (n=227, n=230) | -25.6 (0.91) | -21.4 (0.90)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 6 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-10.5 to -4.2]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 10 data; Test type: Superiority or Other; p = 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.8 to -1.7]

4. Secondary Outcome: Change From Baseline in Mean Trough Diastolic Blood Pressure (22 to 24 Hours After Dosing) as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough diastolic blood pressure measured at each week indicated including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -15.2 (0.70) | -10.6 (0.74)
  Week 10 (n=227; n=230) | -15.1 (0.63) | -12.7 (0.62)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 6 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-6.3 to -2.3]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 10 data; Test type: Superiority or Other; p = 0.006, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.2 to -0.7]

5. Secondary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at each visit indicated including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179, n=162) | -25.7 (0.92) | -19.9 (0.97)
  Week 10 (n=227, n=230) | -26.6 (0.80) | -22.4 (0.79)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 6 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-8.4 to -3.2]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 10 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.4 to -2.0]

6. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at each visit indicated including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -14.7 (0.59) | -10.9 (0.62)
  Week 10 (n=227; n=230) | -15.2 (0.53) | -12.6 (0.53)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 6 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-5.5 to -2.1]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD vs Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate was performed using Week 10 data; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-4.1 to -1.1]

7. Secondary Outcome: Change From Baseline in the Mean Daytime (6 AM to 10 PM) Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at each visit including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -27.0 (0.95) | -20.2 (1.00)
  Week 10 (n=227; n=230) | -27.5 (0.82) | -22.8 (0.82)

8. Secondary Outcome: Change From Baseline in the Mean Daytime (6 AM to 10 PM) Diastolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at each visit including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -15.4 (0.62) | -11.1 (0.65)
  Week 10 (n=227; n=230) | -15.8 (0.55) | -12.9 (0.55)

9. Secondary Outcome: Change From Baseline in the Mean Nighttime (12 AM to 6 AM) Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at each visit indicated including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -21.8 (0.98) | -18.8 (1.03)
  Week 10 (n=227; n=230) | -23.8 (0.87) | -21.1 (0.87)

10. Secondary Outcome: Change From Baseline in the Mean Nighttime (12 AM to 6 AM) Diastolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at each visit indicated including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -12.8 (0.64) | -10.3 (0.67)
  Week 10 (n=227; n=230) | -13.8 (0.60) | -11.9 (0.60)

11. Secondary Outcome: Change From Baseline in the Mean Systolic Blood Pressure at 0 to 12 Hours After Dosing as Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean systolic blood pressure measured at each visit including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -27.7 (0.99) | -20.6 (1.04)
  Week 10 (n=227; n=230) | -28.0 (0.86) | -23.2 (0.86)

12. Secondary Outcome: Change From Baseline in the Mean Diastolic Blood Pressure at 0 to 12 Hours After Dosing as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at each visit including final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline, Week 6 and Week 10.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
mmHg
  Week 6 (n=179; n=162) | -15.7 (0.65) | -11.1 (0.68)
  Week 10 (n=227; n=230) | -16.0 (0.59) | -12.9 (0.58)

13. Secondary Outcome: Percentage of Participants Who Reached Their Trough, Sitting, Clinic Systolic Blood Pressure Targets, Defined as <140 mm Hg for Participants Without Diabetes or Chronic Kidney Disease or <130 mm Hg for Participants With Diabetes or Chronic Kidney Disease
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at each week indicated, defined as <140mm Hg without diabetes or chronic kidney disease or <130/mm Hg with diabetes or chronic kidney disease. Systolic blood pressure is the average of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Week 2, Week 4, Week 6, Week 8 and Week 10.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
percentage of participants
  Week 2 (n=283; n=276) | 33.2 | 34.1
  Week 4 (n=292; n=289) | 68.2 | 54.7
  Week 6 (n=295; n=292) | 71.9 | 58.2
  Week 8 (n=295; n=292) | 79.7 | 65.4
  Week 10 (n=295; n=292) | 76.9 | 69.9

14. Secondary Outcome: Percentage of Participants Who Reached Their Trough, Sitting, Clinic Diastolic Blood Pressure Target, Defined as <90 mm Hg for Participants Without Diabetes or Chronic Kidney Disease or <80 mm Hg for Participants With Diabetes or Chronic Kidney Disease.
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at each week indicated, defined as <90 mm Hg for participants without diabetes or chronic kidney disease or <80 mm Hg for participants with diabetes or chronic kidney disease. Diastolic blood pressure is the average of the 3 serial trough sitting diastolic blood pressure measurements.
Time Frame: Week 2, Week 4, Week 6, Week 8 and Week 10.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
percentage of participants
  Week 2 (n=283; n=276) | 49.1 | 41.3
  Week 4 (n=292; n=289) | 71.9 | 57.4
  Week 6 (n=295; n=292) | 76.6 | 59.2
  Week 8 (n=295; n=292) | 81.4 | 72.3
  Week 10 (n=295; n=292) | 82.7 | 75.0

15. Secondary Outcome: Percentage of Participants Who Reached Their Trough, Sitting, Clinic Systolic and Diastolic Blood Pressure Targets, Defined as <140/90 mm Hg Without Diabetes or Chronic Kidney Disease or <130/80 mm Hg With Diabetes or Chronic Kidney Disease
Description: Percentage of participants who achieve both a clinic systolic and diastolic blood pressure response measured at each week indicated, defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease or <130/80 mm Hg for participants with diabetes or chronic kidney disease[GFR <60 mL/min/1.73 m2 or urinary albumin:creatinine ratio (UACR) >200 mg albumin/g creatinine at Screening.] Systolic/diastolic blood pressure is the average of the 3 serial trough sitting systolic/diastolic blood pressure measurements.
Time Frame: Week 2, Week 4, Week 6, Week 8 and Week 10.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Number analyzed (Participants) | 302 | 303
percentage of participants
  Week 2 (n=283; n=276) | 27.2 | 24.6
  Week 4 (n=292; n=289) | 58.6 | 45.3
  Week 6 (n=295; n=292) | 64.1 | 45.9
  Week 8 (n=295; n=292) | 72.5 | 59.2
  Week 10 (n=295; n=292) | 71.5 | 62.3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD
Serious Adverse Events (participants affected / at risk) | 6/302 | 5/303
Other Adverse Events (participants affected / at risk) | 79/302 | 68/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD (N=302) | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD (N=303)
Angina unstable (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg/Chlorthalidone 12.5 mg QD (N=302) | Azilsartan Medoxomil 40 mg + Hydrochlorothiazide 12.5 mg QD (N=303)
Blood creatinine increased (Investigations) | 38 | 27
Dizziness (Nervous system disorders) | 37 | 32
Headache (Nervous system disorders) | 16 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.